CLINICAL TRIAL: NCT01935258
Title: Psychosomatic Therapy, Feasibility and Cost Analysis, a Pilot Randomised Trial
Brief Title: Psychosomatic Therapy, Feasibility and Cost Analysis
Acronym: PsySom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Tim olde Hartman, Dr T.C. olde Hartman, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/365
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Medically Unexplained Symptoms; Psychosomatic Therapy
Keywords: Medically unexplained symptoms; Somatization; Psychosomatic therapy
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychosomatic therapy (Experimental): Psychosomatic therapy consists of a combination of information and education delivery, relaxation therapy and mindfulness, cognitive approaches and activating therapy. This multi-component approach is captured into a protocol in which therapists are able to modify the treatment in order to deliver a tailor-made treatment for patients with MUS. Psychosomatic therapy delivered by a psychosomatic therapist.
  Interventions: Other: Psychosomatic therapy; Other: care as usual
- care as usual (Other): Usual care of the general practitioner
  Interventions: Other: care as usual

INTERVENTIONS:
Other: Psychosomatic therapy — Psychosomatic therapy delivered by a psychosomatic therapist, consists of a combination of information and education delivery, relaxation therapy and mindfulness, cognitive approaches and activating therapy. This multi-component approach is captured into a protocol in which therapists are able to modify the treatment in order to deliver a tailor-made treatment for patients with MUS.
  Arms: Psychosomatic therapy
Other: care as usual — usual care of the general practitioner

SUMMARY:
Medically unexplained symptoms (MUS) are a common and important problem in primary care. Patients repeatedly presenting MUS to their general practitioner (GP) suffer from their symptoms, are functionally impaired, and are at risk of unnecessary and possibly harmful tests, referrals and treatment. Evidence indicate that specific interventions for patients with MUS, such as reattribution therapy and cognitive behavioural therapy are of limited help. According to experts in this field a multi-component approach is most helpful for these patients.

This pilot trial aims to test the systematic identification of eligible patients, to assess the acceptability of the intervention and to estimate potential treatment effects for a larger trial.

It's a randomised pilot study consisting of patients with MUS in primary care. Patients will be randomized to intervention (usual care and additional psychosomatic therapy) or control condition (usual care alone). Patients will be followed for one year.

Participants are patients consulting their GP more than once with MUS and in which the GP presumes that psychosocial distress is an underlying cause.

The intervention is the psychosomatic therapy delivered by a psychosomatic therapist, consists of a combination of information and education, relaxation therapy and mindfulness, cognitive approaches and activating therapy. This multi-component approach is captured into a protocol in which therapists are able to modify the treatment in order to deliver a tailor-made treatment for patients with MUS.

Primary outcome measures are: the number of patients identified and recruited, perceived symptom severity, measured on a Visual Analogue Scale (VAS) and patients' self-rated symptoms of distress, depression, anxiety and somatization (4DSQ: The Four Dimensional Symptom Questionnaire). Other primary outcome measures are the time needed to include the eligible patients, the number of withdrawals in the intervention and control group, compliance in the therapy group and the number of patients who complete the questionnaires.

Secondary outcome measures are: symptoms of hyperventilation (NHL: Nijmegen Hyperventilation List), physical and mental health status and quality of life (SF-36), and level of functioning (MAF: measure of general functioning). Patient satisfaction with the received therapy is rated on a 5-point Likert-type scale. Medical consumption will be measured by the Cost Diary for medical consumption.

DETAILED DESCRIPTION:
Recruitment and signed informed consent:Participating GPs (n=6) were asked to enrol each consecutive eligible patient and include 10 patients with MUS each. The GPs presented written information and an informed consent form to these patients. Patients had the opportunity to read the information to consider participation before signing the consent form.

Randomisation: Participating patients (n=60) are equally randomised over two groups, the intervention group (usual care and psychosomatic therapy delivered by a psychosomatic therapist) and the control group (usual care of the GP). For the randomisation we used a random number table, whereas a central and blinded allocation procedure was applied.For the randomisation we used a random number table, whereas a central and blinded allocation procedure was applied.

Patients in the intervention group were asked to complete a questionnaire at baseline, at the end of the intervention (+/- 3 months)and at 6 and 12 months. Patients in the control group completed a questionnaire at baseline, at 3 (equals end of intervention), 6 and 12 months.

Statistical analysis The number of patients identified and recruited by the GP as well as the number of eligible patients who declined to enter the trial were analysed using descriptive statistics. Furthermore, at each stage of the study, we recorded the number of trial participants who completed the study.

The effects of the intervention on the primary outcome measures (VAS and 4DSQ) and the secondary outcome measures (NHL, SF-36 and MAF) were estimated using analysis of covariance with baseline value as a covariate. Data analysis was be performed according to the intention-to-treat principle. Medical consumption was measured using the Cost Diary for medical consumption. Patients recorded their absenteeism and healthcare consumption, such as consulting a GP, hospital, paramedic facilities and alternative medicine. Medication intake was recorded at the start and the end of the study. We used standardised Dutch prices (guide cost research 2009), whereas medication costs were calculated according to the Dutch Pharmaco Therapeutic Compass. Costs by absenteeism were calculated according to the Friction Cost method.

Difference in cost of medical consumption between the control and intervention group were estimated using analysis of covariance with baseline value as a covariate.

Difference in baseline characteristics were analysed with the student's t-test for continue variables and the chi-squared test or Fisher's exact test for categorical variables. P-values of < 0.05 were considered statistical significant.

ELIGIBILITY:
Inclusion Criteria:

patients with medical unexplained symptoms who consulting the general practitioner more than once for one or more of the 12 most common symptoms:

* stomach-/abdominal pain,
* back/neck/shoulder pain,
* pain in arms/legs/joints,
* headache, chest pain,
* dizziness,
* fainting spells,
* palpitations of the heart,
* shortness of breath,
* nausea/indigestion,
* feeling tired,
* sleeping disorder and psychosocial distress

Exclusion Criteria:

* patients wich chronic diseases,
* palliative care,
* severe psychiatric disorders,
* long-lasting injury treatment
* patients who are not able to speak, read and write Dutch

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The number of patients identified and recruited | one year
  The number of patients identified and recruited by the GP
The time needed to include the eligible patients | one year
  The time needed to include the eligible patients by the GPs
The number of withdrawals in both groups | one year
  the number of patients that withdraw from the study in both groups
Perceived symptom severity | one year
  Perceived symptoms severity by patients
Patients' self-rated symptoms of distress, depression, anxiety and somatization | one year
  Patients' self-rated symptoms of distress, depression, anxiety ansd somatization measured with the Four Dimensional Symptom Questionnaire (4DSQ)

SECONDARY OUTCOMES:
Symptoms of hyperventilation | at baseline, at 3, 6 and 12 months
  symptoms of hyperventilation measured by the NHL (Nijmegen Hyperventilation List) according to patients
Physical and mental status and quality of life | at baseline, at 3, 6 and 12 months
  Physical and mental health status and quality of life according to patients are measured by the SF-36
Level of functioning | at baseline, at 3, 6 and 12 months
  Level of functioning according to patients are measured by the MAF (measure of general functioning)

OTHER OUTCOMES:
Medical consumption | at baseline, at 3, 6 and 12 months
  Medical consumption will be measured by the Cost Diary for medical consumption.
Baseline characteristics of the participants | at baseline, at 3, 6 and 12 months
  Patient satisfaction with the received therapy is rated on a 5-point Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Tim C. olde Hartman, MD Phd, Principal Investigator — Radboud University Medical Center
Locations (8):
- Netherlands (8):
  - General Practitioner, Douwes Dekker, Albergen, Overijssel
  - General Practitioner, Hesselink, Borne, Overijssel
  - General Practitioner,Tuijnenburg, Enschede, Overijssel
  - General Practitioner, Kleissen, Haaksbergen, Overijssel
  - General Practitioner, van der Waart, Hengelo, Overijssel
  - General Practitioner, Van Rijn, Vriezenveen, Overijssel
  - M. Oijevaar, Borne
  - D.J. Jansen, Julianadorp

REFERENCES:
- [Derived] Wortman MS, Lucassen PL, van Ravesteijn HJ, Bor H, Assendelft PJ, Lucas C, Olde Hartman TC. Brief multimodal psychosomatic therapy in patients with medically unexplained symptoms: feasibility and treatment effects. Fam Pract. 2016 Aug;33(4):346-53. doi: 10.1093/fampra/cmw023. Epub 2016 Apr 13. PMID 27075027